CLINICAL TRIAL: NCT02207023
Title: A Telehealth Intervention to Promote Chronic Disease Management After Stroke: A Pilot Randomized Controlled Study
Brief Title: Healthy Lifestyles After Stroke - Stroke Coach
Acronym: StrokeCoach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Janice Eng, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H13-03353
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Apoplexy; Cerebral Stroke; Cerebrovascular Accident; Cerebrovascular Accident, Acute; Cerebrovascular Apoplexy; Cerebrovascular Stroke; CVA; Stroke, Acute; Vascular Accident, Brain
Keywords: Stroke; Telehealth; Rehabilitation; Stroke Coach; Randomized controlled trial; Lifestyle behaviours; Secondary prevention; Chronic disease self-management
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memory Training Program (No Intervention): Participants will participate in 7 memory training coaching sessions (two in the first month) over a 6 month period. The coaching sessions will be administered by phone.
- Healthy Lifestyle Training Program (Experimental): Participants will participate in 7 lifestyle coaching sessions (two in the first month) over a 6 month period. The coaching sessions will be administered by phone.
  Interventions: Behavioral: Healthy Lifestyle Training Program

INTERVENTIONS:
Behavioral: Healthy Lifestyle Training Program — Study participants in the Healthy Lifestyle Training Program will each receive 7 lifestyle coaching telephone-sessions (30-60 minutes) with a trained lifestyle coach over a 6 month period. The lifestyle coaches will work on a 1:1 basis with each participant to encourage healthy lifestyles.
  Arms: Healthy Lifestyle Training Program

SUMMARY:
The purpose of this study is to examine the efficacy of a lifestyle modification telehealth program on health-related behaviours in community-dwelling individuals living with stroke.

DETAILED DESCRIPTION:
Participants recruited in this study will be randomly assigned to either the Healthy Lifestyle Training Program, or Attention Control Memory Training Program.

Individuals in the Healthy Lifestyle Training Program will each receive 7 lifestyle coaching telephone-sessions (30-60 minutes) with a trained lifestyle coach over a 6 month period. Individuals in the Memory Training Program will each receive 7 memory coaching telephone sessions (30-60 minutes) with a trained memory training coach over a 6 month period. 100 evaluable subjects will be recruited (124 to accommodate for 20% dropout).

ELIGIBILITY:
Inclusion Criteria:

* Has experienced a stroke in the last 12 months
* 50 years of age or older
* Living in the community with phone access
* Mild to moderate stroke severity (i.e., modified Rankin Scale score ranging from 1 to 4)
* Able to communicate in English

Exclusion Criteria:

* Stroke of non-vascular origin
* Actively engaged in formal stroke rehabilitation services
* Uncontrolled arrhythmias
* Significant musculoskeletal or other neurological condition
* Severe aphasia or dysarthria
* Not medically stable
* Pain or co-morbidities which would preclude activity
* Living in long-term residential care
* Cognitive impairment, dependent in activities of daily living, and no caregiver participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-10; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Global measure of lifestyle behavior (Health Promoting Lifestyle Profile II) | End of program (6 months)
  The 52-item Health Promoting Lifestyle Profile II provides a composite score of lifestyle, in the areas of: health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations, and stress management.

SECONDARY OUTCOMES:
Daily walking physical activity | End of program (6 months), and 6 months after the program ends (12 months from baseline)
  Study participants will wear the activity monitor over the 7 days following each assessment period (baseline, 6 months, 12 months)
Dietary behavior (26 items SmartDiet Questionnaire) | End of program (6 months), and 6 months after the program ends (12 months from baseline)
  The SmartDiet Canadian Version Questionnaire was developed to assess fiber and fat intake. This questionnaire has 26 questions about diet and lifestyle. Most questions list foods in 3 or 4 categories according to fat or fiber content.
Medication adherence (8-item Morisky Medication Adherence Scale) | End of program (6 months), and 6 months after the program ends (12 months from baseline)
  The Morisky Medication Adherence Scale assesses habits in taking medication and barriers that may hinder medication adherence.
Depressive symptoms (20-item Centre for Epidemiological Studies-Depression [CES-D] Scale) | End of program (6 months), and 6 months after the program ends (12 months from baseline)
  This scale assess the frequency with which participants experience depression symptoms, such as restless sleep, poor appetite, and feeling lonely, during the past week.
Cognition (Montreal Cognitive Assessment [MoCA]) | End of program (6 months), and 6 months after the program ends (12 months from baseline)
  The MoCA is a screening instrument to assess for cognitive impairment.
Cardiovascular risk factors (resting blood pressure, lipid, and glucose profiles, C-Reactive Protein, Homocysteine). | End of program (6 months), and 6 months after the program ends (12 months from baseline)
  These risk factors will be assessed using hospital lab services.
Body composition (Body Mass Index, waist circumference) | End of program (6 months), and 6 months after the program ends (12 months from baseline)
  The Body Mass Index is a measure of body fat based on weight and height. Waist circumference will be measured using a tape measure around the waist at the height of the umbilicus.
Health-related quality of life (SF-36) | End of program (6 months), and 6 months after the program ends (12 months from baseline)
  The SF-36 is a generic health status measure that was designed to be applied to all health conditions and assess health concepts, which represent basic human values and are relevant to a person's functional status and well-being.
Health and Social Services Utilization (Health and Social Service Utilization Inventory) | End of program (6 months), and 6 months after the program ends (12 months from baseline)
  The Health and Social Services Utilization inventory collects data regarding health services used, medications, and out of pocket health costs.
Global measure of lifestyle behavior (Health Promoting Lifestyle Profile II) | 6 months after the program ends (12 months from baseline)
  The 52-item Health Promoting Lifestyle Profile II provides a composite score of lifestyle, in the areas of: health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations, and stress management.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Eng, PhD, Principal Investigator — University of British Columbia
Locations (7):
- Canada (7):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - University Hospital of Northern BC, Prince George, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Holy Family Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - GF Strong Rehabilitation Centre, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakakibara BM, Lear SA, Barr SI, Goldsmith CH, Schneeberg A, Silverberg ND, Yao J, Eng JJ. Telehealth coaching to improve self-management for secondary prevention after stroke: A randomized controlled trial of Stroke Coach. Int J Stroke. 2022 Apr;17(4):455-464. doi: 10.1177/17474930211017699. Epub 2021 May 27. PMID 33949270
- [Derived] Sakakibara BM, Lear SA, Barr SI, Benavente O, Goldsmith CH, Silverberg ND, Yao J, Eng JJ. A telehealth intervention to promote healthy lifestyles after stroke: The Stroke Coach protocol. Int J Stroke. 2018 Feb;13(2):217-222. doi: 10.1177/1747493017729266. Epub 2017 Sep 4. PMID 28869405